CLINICAL TRIAL: NCT02689466
Title: Cholinergic Receptor Imaging in Dystonia
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160064; 16-N-0064
Record Dates: First submitted 2016-02-20; First posted 2016-02-24 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2025-10-03

CONDITIONS: Cervical Dystonia; Dystonia; Movement Disorder; Focal Dystonia
Keywords: Adult; Acetylcholine; Movement Disorder; Magnetic Resonance Imaging (MRI); PET Imaging; Natural History
MeSH Terms: conditions — Torticollis; Dystonia; Movement Disorders; Dystonic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cervical dystonia: clinically documented cervical dystonia (focal cervical or segmental with neck involvement) established by history and physical/neurological examination, at least 18 years old.
  Interventions: Drug: [18F]FP-TZTP
- healthy volunteers: age and sex matched healthy volunteers, at least 18 years old.
  Interventions: Drug: [18F]FP-TZTP

INTERVENTIONS:
Drug: [18F]FP-TZTP — radioligand

SUMMARY:
Background:

Dystonia is a movement disorder in which a person s muscles contract on their own. This causes different parts of the body to twist or turn. The cause of this movement is unknown. Researchers think it may have to do with a chemical called acetylcholine. They want to learn more about why acetylcholine in the brain doesn t work properly in people with dystonia.

Objective:

To better understand how certain parts of the brain take up acetylcholine in people with dystonia.

Eligibility:

Adults at least 18 years old who have DYT1 dystonia or cervical dystonia.

Healthy adult volunteers.

Design:

Participants will be screened with a medical history, physical exam, and pregnancy test.

Study visit 1:

Participants will have a magnetic resonance imaging (MRI) scan of the brain. The MRI scanner is a metal cylinder in a strong magnetic field that takes pictures of the brain. Participants will lie on a table that slides in and out of the cylinder.

Study visit 2:

Participants will have a positron emission tomography (PET) scan. The PET scanner is shaped like a doughnut. Participants will lie on a bed that slides in and out of the scanner. A small amount of a radioactive chemical that can be detected by the PET scanner will be given through an IV line to measure how the brain takes up acetylcholine.

...

DETAILED DESCRIPTION:
Dystonia is a heterogeneous group of movement disorders characterized by abnormal muscle contractions resulting in abnormal postures and movements. The spectrum of dystonia includes focal, segmental, multifocal, and generalized presentations with a broad range of age of onset. An example of a focal dystonia is cervical dystonia. The pathophysiology of dystonia is unclear, but prior neuroimaging and neuropathological studies have identified a role for the basal ganglia. In neuroimaging studies, microstructural changes in the basal ganglia have been found in voxel based morphometry (VBM) and diffusion tensor imaging (DTI), and abnormal basal ganglia metabolism has been seen in imaging with fluorodeoxyglucose positron emission tomography (FDG-PET) in various types of dystonia. Basal ganglia pathology has been observed, including a case series reporting neuronal loss in the striatum. There is further evidence implicating the basal ganglia in dystonia from studies of animal models. In animal models, experimental lesions of the basal ganglia induced dystonia. An abnormality in cholinergic neurotransmission has been has also been suggested because of a clinical response to antimuscarinic medications. The striatum is a site of acetylcholine synthesis, and expresses muscarinic receptors. While antimuscarinic medications are useful in the symptomatic treatment of dystonia, the role of muscarinic acetylcholine neurotransmission in dystonia is unclear.

Objective

The objective of this application is to determine the role played by a major basal ganglia neurotransmitter, acetylcholine, in the pathophysiology of primary dystonia. The central hypothesis is that cholinergic neurotransmission is deficient in the striatum in dystonia.

Study Population

We plan to examine one group of patients with a form of primary dystonia (cervical dystonia) to be compared with healthy volunteers without history of neurological or major psychiatric disorders (stable mild anxiety or stable mild depression are allowed).

Design

This is a case-control study. Using a neuroimaging technique, position emission tomography (PET), the central hypothesis will be tested by pursuing one specific aim: to map M2 muscarinic acetylcholine receptor binding in cervical dystonia as measured with PET using [18F]FP-TZTP.

Outcome Measures

This study will determine cholinergic neurotransmitter receptor binding in patients with cervical dystonia compared with healthy controls. This proposed research study is expected to advance our understanding of the pathophysiology of dystonia in order to identify possible targets for potential pharmacological treatments in dystonia and monitor disease progression.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy research volunteers and adult patients with cervical dystonia will be eligible for the study.

1. Adult patients with cervical dystonia will have clinically documented cervical dystonia (focal cervical or segmental with neck involvement)established by history and physical/neurological examination.

   --Cervical dystonia patients must not have had received botulinum toxin injections into neck muscles for at least about 10 weeks at time of study participation
2. Healthy volunteers will be healthy subjects without neurological or psychiatric disorders (except for stable mild anxiety or stable mild depression) established by history and physical/neurological examination.
3. All participants will be at least 18 years of age. There is no maximum age limit.
4. Participants must be able to abstain from tobacco or nicotine replacement for at least 3 days prior to PET scan if participating in both MRI and PET scanning..
5. Participants must be able to abstain from caffeine for at least 24 hours prior to PET scan if participating in both MRI and PET scanning.
6. Participants must be able to fast for 3 hours before PET scan if participanting in both MRI and PET scanning.

EXCLUSION CRITERIA:

1. Subjects who are incapable of giving informed consent.
2. Employees of NINDS
3. Pregnant or breastfeeding women. Aside from history obtained at the screening, pregnancy status in women with childbearing potential is also established by urine pregnancy testing no more than 24 hours before each MRI and PET scan session.
4. Subjects with past or present medical history of (a) neurological disorders, such as stroke, movement disorders (other than cervical dystonia in the patient group), brain tumors, traumatic brain injury with loss of consciousness lasting more than a few seconds, ataxias, myopathies, myasthenia gravis, demyelinating diseases, alcoholism, drug dependence; (b) psychiatric disorders besides stable mild anxiety or stable mild depression, such as schizophrenia, major depressive and/or bipolar disorder, obsessive-compulsive disorder; (c) ventricular arrhythmias, renal and hepatic insufficiency, vascular headache, or carcinoid syndrome.
5. Abnormalities in neurological examination other what is typically associated with cervical dystonia, or any abnormalities in neurological examination in healthy volunteers.
6. Subjects who are currently taking oral medications known to affect muscarinic acetylcholine receptor binding in the central nervous system. Of note, some over-the counter-medications are known to affect muscarinic acetylcholine receptor binding. Subjects who use medications known to affect muscarinic acetylcholine receptor binding, such as first generation antihistamines for common cold and allergy symptoms and sleep aids for insomnia, occasionally on an as needed basis may be enrolled in this study. Furthermore, these as needed medications should be paused for at least 3 days before PET scanning. This three-day period is equivalent to about 4 to 5 half lives for these medications. In addition, subjects who use topical antimuscarinic medications, such as eye drops for glaucoma and inhalers, may be enrolled in this study because topical antimuscarinic medications have negligible systemic bioavailability. Subjects who have contraindications to MRI, ferromagnetic objects in their bodies (e.g., implanted stimulators including deep brain stimulation, aneurysm clips, prosthesis, artificial heart valves, etc.) that cannot be removed for the purpose of study participation.
7. Subjects who have claustrophobia.
8. Subjects who are unable to lie comfortably on their back for about one hour for MRI scanning (and about two hours for PET scanning if participating in both MRI and PET scanning).
9. Subjects with any radiation exposure in the past year that, together with the research PET scan, would exceed the NIH Radiation Safety Committee s annual limit (5 rem) if participating in both MRI and PET scanning.
10. Cervical dystonia patients who have cervical dystonia associated with trauma

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the pool of former participants in the studies of the Human Motor Control Section including but not limited to Protocol 93-N-0202 ( Diagnosis and Natural History Protocol for Patients with Different Neurological Conditions ), through the Healthy Volunteer and Patient Recruitment Office at NIH, advertisements in Dystonia Medical Research Foundation (DMRF) and Tyler s Hope organization newsletters and on their websites, and through contacts with referring physicians following approval of this protocol. Employees of the NINDS will not be recruited, but employees of the other NIH institutes may participate.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Characterize the M2 muscarinic acetylcholine receptor binding in DYT1 dystonia and cervical dystonia patients as measured with high-resolution positron emission tomography (PET) using [18F]FP-TZTP. | throughout protocol
  Characterization of the M2 muscarinic acetylcholine receptor binding in cervical dystonia patients as measured with high-resolution PET using [18F]FP-TZTP.

CONTACTS AND LOCATIONS:
Overall Officials: Silvina G Horovitz, Ph.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-N-0064.html